CLINICAL TRIAL: NCT05338619
Title: A Phase II, Multicenter Study of Lazertinib as Consolidation Therapy in Patients With Locally Advanced, Unresectable, EGFR Mutation Positive Non-Small Cell Lung Cancer (Stage III) Who Have Not Progressed Following Definitive, Platinum-based, Chemoradiation Therapy (PLATINUM Trial)
Brief Title: A Study of Lazertinib as Consolidation Therapy in Patients With Locally Advanced, Unresectable, EGFR-Mutant Non-Small Cell Lung Cancer (Stage III) Following Chemoradiation Therapy
Acronym: PLATINUM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sung Yong Lee (Other)
Collaborators: Yuhan Corporation (Industry)
Responsible Party: Sponsor-Investigator, Sung Yong Lee, Professor, Korea University Guro Hospital
Organization: Korea University Guro Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Korea-Lazertinib-CCRT; LASER IIT-010 (Other Grant/Funding Number: YUHAN Coorporation)
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer Stage III; EGFR Positive Non-small Cell Lung Cancer; Non-squamous Non-small-cell Lung Cancer
Keywords: NSCLC; Non-squamous cell carcinoma; EGFR; EGFR-TKI; Lazertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib

STUDY DESIGN:
Intervention Model Description: Lazertinib treatment group (open-label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lazertinib (Experimental): Lazertinib 240mg, oral, QD
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib — Lazertinib 240mg (3 Tabs as Laclaza Tab 80mg) once daily in oral can continue until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Other Names: LECLAZA

SUMMARY:
The "PACIFIC" trial confirmed that the consolidation therapy with durvalumab in patients with stage III, locally advanced, unresectable NSCLC that had not progressed after definitive platinum-based chemoradiation therapy improved the progression-free survival (PFS) by about 17 months. However, in PACIFIC, no significant differences between durvalumab and placebo were observed in PFS. Unmet need remains in development of successful consolidation therapy following chemoradiation therapy in patients with EGFR-mutant stage III unresectable NSCLC.

A recent "ADAURA" study showed that Osimertinib as an adjuvant therapy after surgery significantly prolonged disease-free survival in EGFR mutation-positive patients. Lazertinib, like Osimertinib, is a third-generation EGFR TKI agent and has shown excellent anticancer effects in preclinical studies and in early clinical settings. Based on these results of the 3rd generation EGFR TKI, Lazertinib, it is expected that there is a clinical benefit Lazertinib as consolidation therapy.

This study aims to investigate the clinical benefits of Lazertinib (Trade name: LECLAZA Tab) consolidation therapy for patients with EGFR mutation-positive, unresectable stage III NSCLC after definitive platinum-based chemoradiation therapy.

DETAILED DESCRIPTION:
This study is designed as a prospective, open-label, single-arm, multicenter, phase II, investigator-initiated trial. A total of 77 patients will participate in the study who have undergone definitive platinum-based concurrent chemoradiation therapy and have no disease progression. Patients are to be enrolled within 1 to 42 days after concurrent chemoradiation therapy and to be administrated with lazertinib 240mg oral once daily until disease progression, or unacceptable toxicity. Patients will visit every 8 weeks and perform CT/MRI tumor evaluation by investigator, and will be followed up for survival every 3 months by phone thereafter. Patients will be followed up till maximum of appropriately 4 years of which 3 years since the last patient enrollment must be.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older
2. Histologically and cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC) non-squamous cell carcinoma who present with locally advanced, unresectable, Stage III disease
3. ECOG PS 0,1
4. Expected life expectancy of 6 months and more
5. Patients who have received at least 2 cycles of definitive platinum-based concurrent chemoradiation therapy (CCRT) and who must be within 1 to 42 days after completion of radiation therapy
6. Patients must not have had disease progression during or following CCRT
7. Patients with adequate organ and bone marrow function
8. Patients who give in written consent voluntarily to participate in this study

Exclusion Criteria:

1. History of interstitial lung disease, drug-induced interstitial lung disease, or radiation interstitial pneumonia
2. History of other primary malignancy
3. Mixed small cell and NSCLC histology
4. Prior treatment with EGFR-TKI Therapy
5. Unresolved toxicity of CTCAE grade 2 or higher following chemoradiation
6. Current history of CTCAE grade 2 or higher pneumonia prior to chemoradiation therapy
7. Patients with severe hypersensitivity to active ingredient or excipient of the investigational medicinal product
8. Pregnant or breastfeeding patients
9. Patients who do not agree to contraception with medically acceptable method for at least 6 months after the end of study intervention treatment
10. Patients who participated in clinical trials within 4 weeks before participating in this study
11. Judgment by the investigator that the patient is unsuitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Tumor scan will be performed at baseline the every 8 weeks until confirmed disease progression (up to 4 years)
  The time from the date of enrollment until the date of disease progression or death (by any cause in the absence of progression) Per RECIST 1.1 as assessed by Investigator.

SECONDARY OUTCOMES:
Overall survival (OS) | Until death (up to maximum of approximately 4 years)
  The time from the date of enrollment until the date of death
Objective response rate (ORR) | Tumor scan will be performed at baseline the every 8 weeks until confirmed disease progression (up to 4 years)
  The number (%) of patient at least 1 visit response of Complete response (CR) or Partial response (PR).
  Per RECIST 1.1 as assessed by Investigator.
Duration of response (DoR) Duration of response (DoR) | Tumor scan will be performed at baseline the every 8 weeks until confirmed disease progression (up to 4 years)
  The time from the date of first documented response until the first date of documented progression (or death in the absence of disease progression) Per RECIST 1.1 as assessed by Investigator.
Time to death or distant metastasis (TTDM) | Until death or distant metastasis (up to maximum of approximately 4 years)
  The time from the date of enrollment until the first date of distant metastasis or death in the absence of distant metastasis.
  Per RECIST 1.1 as assessed by Investigator.
Safety profile : Adverse Events according to CTCAE V5.0 | every visit (up to maximum of approximately 4 years)
  Adverse events, Serious adverse events or other significant safety findings

OTHER OUTCOMES:
Changes form baseline in different biomarkers | Pre-dose(within 6 week of completion of CCRT), after 8-week dosing, and confirmed disease progression (approximately 15 months)
  Biomarker evaluations include tumor-educated platelets (TFP), circulating tumor DNA(ctDNA), and peripheral blood mononuclear cells (PMBCs).
  It will be investigated to understand the better and long-term survival, drug-resistant mechanism and hematology in occurrence of pneumonitis.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Lee, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (13):
- South Korea (13):
  - Kosin University Gospel Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital Hwasun Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Koera University Guro Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi J, Lee JE, Choi CM, Oh IJ, Lee KY, Jang TW, Lee SH, Kim EY, Park DW, Park SH, Lee SY. A phase II, multicenter study of lazertinib as consolidation therapy in patients with locally advanced, unresectable, EGFR mutation-positive non-small cell lung cancer (stage III) who have not progressed following definitive, platinum-based, chemoradiation therapy (PLATINUM trial). Thorac Cancer. 2022 Dec;13(23):3431-3435. doi: 10.1111/1759-7714.14663. Epub 2022 Oct 19. PMID 36259253
- [Derived] Wang W, Wang Q, Xu C, Li Z, Song Z, Zhang Y, Cai X, Zhang S, Lian B, Li W, Liu A, Zhan P, Liu H, Lv T, Miao L, Min L, Chen Y, Yuan J, Wang F, Jiang Z, Lin G, Pu X, Rao C, Lv D, Yu Z, Li X, Tang C, Zhou C, Xie C, Zhang J, Guo H, Chu Q, Meng R, Wu J, Zhang R, Wang L, Zhu Y, Hu X, Xie Y, Lin X, Cai J, Lan F, Feng H, Wang L, Yao W, Shi X, Huang J, Chen H, Zhang Y, Sun P, Wan B, Pang F, Xu Z, Wang K, Xia Y, Ye M, Wang D, Wei Q, Feng S, Zhou J, Zhang J, Lv D, Gao W, Kang J, Yu G, Liang X, Yu C, Shi L, Yang N, Wu L, Hong Z, Hong W, Fang M, Zhang Y, Lu Y, Wang G, Ma S, Si L, Fang W, Song Y. Chinese expert consensus on the multidisciplinary management of pneumonitis associated with immune checkpoint inhibitor. Thorac Cancer. 2022 Dec;13(23):3420-3430. doi: 10.1111/1759-7714.14693. Epub 2022 Oct 21. PMID 36268845